CLINICAL TRIAL: NCT01974908
Title: Using Fibrillatory Factor to Predict the Source of Ventricular Tachycardia in Man
Brief Title: Fibrillatory Factor in Ventricular Tachycardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Jaswinder Gill, M.D., Consultant Electrophysiologist and Professor of Cardiology, Guy's and St Thomas' NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GSTT-FF-1
Record Dates: First submitted 2013-07-13; First posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ventricular Tachycardia (VT) (Experimental): Patients with VT will undergo a clinically indicated ablation of their VT
  Interventions: Procedure: Fibrillatory Factor calculation (FF)

INTERVENTIONS:
Procedure: Fibrillatory Factor calculation (FF) — During sinus rhythm these patients will undergo a simple pacing protocol to allow us to calculate FF, which is an area we would predict is mod likely to be the origin of their VT.

SUMMARY:
This study involves recording electrical signals inside the heart during an ablation procedure. It is thought that by studying these electrical signals in detail the investigators may be able to better identify and treat patients at risk of Ventricular Tachycardia (VT).

VT is where the lower chambers (ventricles) of your heart beat fast and this condition can be life-threatening. An ablation procedure is performed in patients who have VT despite the best treatment available with tablets.

Cardiac ablation involves interrupting the abnormal electrical signals, which cause VT, by applying a type of electrical energy through a catheter. An important part of the ablation procedure is the identification of the exact part of the heart muscle responsible for causing the VT. This typically involves sampling the electrical signals in lots of different areas of the heart, which allows the construction of computer generated 3 dimensional pictures of the structure and the electrical circuits inside the ventricle. Recent research has identified a new method to interpret these electrical signals (called Fibrillatory Factor - FF), which may allow better identification of the area within the ventricle that should be ablated.

A standard VT ablation will often involve us controlling the heart-beat by pacing the heart through 1 of the investigators catheters within the heart. The electrical response to pacing at different heart rates can often provide your doctor with information to help the ablation. This study will involve an additional period of pacing at different heart rates, during which the electrical response is measured in different areas around the ventricle. This will allow us to calculate areas of the ventricle, which the investigators new measure FF would predict to be the source of the VT. In the future this may then allow us to better identify patients who are at risk of VT, and to better locate the area that needs to be ablated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above, and capable of giving informed consent
* Scheduled for a clinically indicated cardiac ablation for the treatment of ventricular tachycardia

Exclusion Criteria:

* Moderate or severe aortic stenosis or mitral stenosis
* Active infection
* Presence of thrombus, cardiac tumour, interatrial Baffle patch (a specific form of congenital cardiac surgery) or prior septal occluder device
* Subjects who cannot be anticoagulated of infused with heparinized saline
* A history of heparin induced thrombocytopenia
* Pregnant or actively breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Fibrillatory Factor | 18 months
  To identify the proportion of clinical VT circuits which could be predicted during sinus rhythm from the calculation of fibrillation factor. The number of FF derived VT exit points which are successfully predicted blindly by the investigators (using the clinically derived VT exit point based on electrophysiology assessment and ablation) will be the primary endpoint.

SECONDARY OUTCOMES:
Real-time fibrillatory factor | 18 months
  Having established that fibrillatory factor (FF) can predict VT circuits we will then develop our software further so that we can calculate FF in real-time. This will then be used in further research studies to guide invasive mapping.

CONTACTS AND LOCATIONS:
Overall Officials: Jaswinder Gill, MD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guys and St Thomas' NHS Trust, London, United Kingdom